CLINICAL TRIAL: NCT05836870
Title: Tele-PancFit: A Multi-site Trial of Video-based Strengthening Exercise Prehabilitation for Patients With Resectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0033; NCI-2023-03448 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A-Enhanced Usual Care (Experimental): Participants will be given general recommendations to increase physical activity and improve nutrition before surgery.
  Interventions: Other: Enhanced Usual Care
- Group B-Tele-supervised resistance exercises (Experimental): Participants will take part in a monitored exercise program. The study team will provide more instructions and information about the program
  Interventions: Behavioral: Tele-supervised resistance exercises

INTERVENTIONS:
Other: Enhanced Usual Care — Participants will receive general recommendations to maintain physical activity.
  Arms: Group A-Enhanced Usual Care
Behavioral: Tele-supervised resistance exercises — Participants will take part in a monitored exercise program.
  Arms: Group B-Tele-supervised resistance exercises

SUMMARY:
To learn if a supervised exercise program during chemotherapy treatments can help to improve outcomes in patients who have been diagnosed with pancreatic cancer

DETAILED DESCRIPTION:
Primary Objectives:

Compare the rate of adjuvant chemotherapy initiation in patients who receive Tele-PancFit (telesupervised strengthening and remotely-monitored moderate intensity aerobic exercise) versus an enhanced usual care group who receive general recommendations for physical activity and receive an activity tracker.

Hypothesis: Tele-PancFit participation (Arm B) will improve the rate of adjuvant therapy compared to enhanced usual care (Arm A).

Secondary Objectives:

1. Determine the effects of Tele-PancFit intervention on HRQOL among patients with localized PDAC, including the change of the HRQOL over time and the between study groups.
2. Compare skeletal muscle maintenance indicated by SMI using CT between patients in the exercise and UC groups of the Tele-PancFit intervention.
3. Define the effects of Tele-PancFit participation on tumor vascular density and maturity among patients undergoing neoadjuvant chemotherapy for PDAC.

   Other exploratory objectives include:
4. Determine the effects of the Tele-PancFit intervention on secondary physical function, symptom and body composition study measures. Compare changes between baseline, preoperative and postoperative timepoints within each study arm and between study arms of the following measures. Also compare outcome values between study arms at each data collection timepoint.

   1. Skeletal muscle maintenance (skeletal muscle index [SMI] using routinely-obtained CT scans)
   2. Skeletal muscle quality (skeletal muscle density [SMD] using routinely-obtained CT scans)
   3. Visceral fat and subcutaneous fat using routinely-obtained CT scans
   4. Muscle strength (1-RM chest press,1-RM leg press, 30 second chair stand test and 30 second arm curl test)
   5. Muscle endurance
   6. Submaximal exercise capacity (6MWT)
   7. Self-reported exercise (Modified Godin)
   8. Self-reported physical functioning (PROMIS Cancer Function)
   9. Fatigue (FACIT-F)
   10. HRQOL (FACT-Hep)
5. To compare levels of circulating tumor-associated and angiogenic factors such as CA 19-9, thrombospondin, CXCL12, IL-1b, VEGF, S1P between groups upon enrollment (T0), following administration of preoperative therapy (T1), and at postoperative visits (T2a/b).
6. To compare cancer associated fibroblasts (CAFs), and tumor infiltrating immune cells between groups (among patients who have undergone surgical resection).
7. Determine the effects of the Tele-PancFit intervention on oncology treatment outcomes by comparing these measures in the Arms A and B:

   1. Completion of intended NT dose
   2. Dose reduction or change in NT treatment plan
   3. Time of initiation of AT after surgery
   4. Dose reduction or change in AT treatment plan
   5. Completion of AT (6 months total perioperative chemotherapy)
   6. incidence of perioperative adverse events that occur within 90 days between groups (Accordion score)
   7. Hospital length of stay
   8. Acute cancer care center or emergency center visits within 30 days of surgery
8. Evaluate the effects of adherence to nutritional recommendations to body composition and physical function. Evaluate the effects of weight loss and sarcopenia status (yes/no) on body composition.
9. To assess the change in nutrition status (PGSGAsf) along all study time points in all enrolled participants. Also, to correlate the PGSGAsf score with the corresponding anthropometric measures at each time point for all participants.
10. To examine differences among Fitbit-measured physical activity and sleep between groups and associations among Fitbit variables and secondary endpoints between and within groups.
11. To compare the 6MWT distance and secondary endpoints of participants within subgroups of patients who are stratified as "active" versus "insufficiently active" based on the Godin-Shephard Leisure Time Physical Activity Questionnaire.
12. To compare the 6MWT distance and secondary endpoints of participants within subgroups of patients with different levels of physical activity (light, moderate, high intensity activity).
13. To explore the effect of sociodemographic variables (sex, age, race/ethnicity, zip code [for urban vs rural classification], distance form the hospital, marital status, insurance), need to borrow devices and Wi-Fi connection on patient clinical outcomes and adherence to the activity prescription.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form
* Biopsy-proven pancreatic adenocarcinoma, resectable/borderline resectable (T1-3, N0-2, M0)
* Recommended to receive 2-6 months of neoadjuvant chemotherapy followed by surgical resection including participants who have not yet received chemotherapy and participants who have already received their first cycle of chemotherapy.
* Willingness to adhere to the Tele-PancFit study intervention
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Able to schedule baseline (T0) appointment for fitness testing and program teaching at the fitness testing location at each study site or able to schedule remote fitness testing and program teaching:

  1. Behavioral Research and Treatment Center (BRTC) at MDACC
  2. Exercise Physiology laboratory in the Department of Kinesiology and Health Education at UT Austin
  3. Outpatient Rehabilitation gymnasium at Banner MDA
* Able to understand the description of the study, exercise program, and willing to participate
* Home or community access to wireless internet (Wi-Fi) and agreement to engage with study personnel for real-time tele-RT sessions
* Age ≥ 18
* Meet all screening requirements (described below).

Exclusion criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Non-English speaking
* Has participated in regular RT (RT for all major muscle groups at least twice per week) throughout the month prior to recruitment
* Unable to complete the baseline assessment questionnaires or functional assessments
* Screen failure for exercise safety based on PAR-Q and/or PROMIS questions as described in section 4.4 (Screening Procedure).
* Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease (New York Heart Association functional class III or IV).
* Recent fracture or acute musculoskeletal injury that precludes the ability to weight bear fully on all 4 limbs in order to participate in an exercise intervention.
* Numeric pain rating scale of ≥7 out of 10
* Myopathic or rheumatologic disease that impacts physical function.
* (Females only) Known pregnancy, as communicated to study personnel by clinicians in GI Medical Oncology; females of childbearing potential receive advice to use methods of contraception per usual care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | thorugh study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: An Ngo-Huang, DO, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org